CLINICAL TRIAL: NCT00400569
Title: Phase II Open-Label Study of Sunitinib Malate (SU011248) in Adult Patients With Metastatic and/or Surgically Unresectable Soft Tissue Sarcoma
Brief Title: Phase II Study of Sunitinib Malate for Metastatic and/or Surgically Unresectable Soft Tissue Sarcoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MCC-14902; GA618075 (Other: Pfizer Pharamaceutic)
Record Dates: First submitted 2006-11-15; First posted 2006-11-17 (Estimated); Results first posted 2012-08-28 (Estimated); Last update posted 2012-08-28 (Estimated); Status verified 2012-07

CONDITIONS: Liposarcoma; Leiomyosarcoma; Fibrosarcoma; Malignant Fibrous Histiocytoma
Keywords: Sunitinib malate; SUTENT; SU011248; Soft tissue sarcoma; Gastrointestinal stromal tumors (GIST); MFH; Tyrosine kinase inhibitor; Imatinib mesylate; Phase II
MeSH Terms: conditions — Liposarcoma; Leiomyosarcoma; Fibrosarcoma; Histiocytoma, Malignant Fibrous; Sarcoma; Gastrointestinal Stromal Tumors | interventions — Sunitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Sunitinib Malate (SU011248) Treatment (Experimental): Sunitinib malate, 50 mg daily, for 4 weeks every 6 weeks
  Interventions: Drug: Sunitinib Malate (SU011248)

INTERVENTIONS:
Drug: Sunitinib Malate (SU011248) — For each 6 week cycle, patients will take SU011248 every day in the morning for 4 weeks followed by a 2 week rest period.
  Other Names: Sutent; SU011248

SUMMARY:
This is an open label single site Phase II clinical trial to identify a potentially promising therapy dose for Sunitinib malate. The study drug will be taken orally once daily on days 1 through 28 of each 42 day cycle. Treatment will be continued until there is either disease progression or cumulative/acute toxicity.

All patients with unresectable or metastatic soft tissue sarcoma (STS): leiomyosarcoma, liposarcoma, fibrosarcoma, and malignant fibrous histiocytoma (MFH) seen at the Moffitt Cancer Center will be screened for eligibility to be enrolled in the study.

DETAILED DESCRIPTION:
This is an open label single site Phase II clinical trial to identify a potentially promising therapy dose for Sunitinib malate, an oral multi-kinase inhibitor. The study drug will be taken orally once daily on days 1 through 28 of each 42 day cycle. Treatment will be continued until there is either disease progression or cumulative/acute toxicity which in the opinion of the treating physician or the trial Principal Investigator (PI) compromises the ability of the patient to receive treatment or the patient desires to stop treatment.

All patients with unresectable or metastatic STS: leiomyosarcoma, liposarcoma, fibrosarcoma, and MFH seen at the Moffitt Cancer Center will be screened for eligibility to be enrolled in the study.

An office visit will be required before the beginning of every cycle every 6 weeks to assess toxicity and for physical examination. Complete blood count (CBC) and differential, comprehensive metabolic panel, and electrocardiogram (ECG) will be obtained at every scheduled visit.

ELIGIBILITY:
Inclusion Criteria:

* Resolution of all acute toxic effects of prior chemotherapy or radiotherapy or surgical procedures to National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) Version 3.0 grade less than or equal to 1.
* Adequate organ function as defined by the following criteria:

  * Serum aspartate transaminase (AST) and serum alanine transaminase (ALT) less than or equal to 2.5 x local laboratory upper limit of normal (ULN), or AST and ALT less than or equal to 5 x ULN if liver function abnormalities are due to underlying malignancy
  * Total serum bilirubin less than or equal to 1.5 x ULN
  * Absolute neutrophil count (ANC) greater than or equal to1500/microL
  * Platelets greater than or equal to 100,000/microL
  * Hemoglobin greater than or equal to 9.0 g/dL
  * Serum calcium less than or equal to 12.0 mg/dL
  * Serum creatinine less than or equal to 1.5 x ULN
* Histologically-proven liposarcoma, leiomyosarcoma, fibrosarcoma, or MFH
* Measurable disease radiographically
* Disease that is deemed surgically unresectable and/or metastatic
* Age greater than or equal to 18 years
* Life expectancy greater than 16 weeks
* Eastern Cooperative Oncology Group (ECOG) performance status less than or equal to 2
* Patients may have had up to 3 prior chemotherapies within 4 weeks of starting the study treatment.

Exclusion Criteria:

* Major surgery or radiation therapy or chemotherapy within 4 weeks of starting the study treatment.
* NCI CTCAE version 3 grade 3 hemorrhage within 4 weeks of starting the study treatment.
* History of or known brain metastases, spinal cord compression, or carcinomatous meningitis, or evidence of symptomatic brain or leptomeningeal disease.
* Any of the following within the 6 months prior to study drug administration:

  * myocardial infarction,
  * severe/unstable angina,
  * coronary/peripheral artery bypass graft,
  * symptomatic congestive heart failure,
  * cerebrovascular accident or transient ischemic attack, or pulmonary embolism
* Ongoing cardiac dysrhythmias of NCI CTCAE greater than or equal to grade 2
* Prolonged QTc interval on baseline electrocardiogram (ECG) > 500 msec.
* Hypertension that cannot be controlled by medications (>150/100 mm Hg despite optimal medical therapy)
* Prior tyrosine kinase inhibitor therapy
* Pre-existing thyroid abnormality with thyroid function that cannot be maintained in the normal range with medication
* Known human immunodeficiency virus (HIV) or acquired immunodeficiency syndrome (AIDS)-related illness or other active infection
* Concurrent treatment on another clinical trial, except supportive care or non-treatment trials
* Concomitant use of agents known to induce or inhibit CYP3A4
* Concomitant use of agents metabolized by the cytochrome P450 system
* Ongoing treatment with therapeutic doses of Coumadin (low dose Coumadin up to 2 mg by mouth [PO] daily for thrombo-prophylaxis is allowed)
* Pregnancy or breastfeeding patients
* Other severe acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or study drug administration, or may interfere with the interpretation of study results, and in the judgment of the investigator would make the subject inappropriate for entry into this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2006-11; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alberto Chiappori, M.D., Principal Investigator — H. Lee Moffitt Cancer Center and Research Institute
Locations (1):
- H. Lee Moffitt Cancer Center & Research Institute, Tampa, Florida, United States

REFERENCES:
- See also: Moffitt Cancer Center Clinical Trials Website — http://www.moffitt.org/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: From September 2006 to August 2007, a total of 48 patients were enrolled on the study by the Moffitt Cancer Center Sarcoma Program. In general, the patients had been heavily pretreated previously, with a significant number receiving more than one prior chemotherapy regimen and most with multiple metastatic sites.
Groups:
- Experimental: Sunitinib Malate (SU011248) Treatment: Sunitinib malate, 50 mg daily, for 4 weeks every 6 weeks
Period: Overall Study
Arm/Group | Experimental: Sunitinib Malate (SU011248) Treatment
Started | 48
Completed | 47
Not Completed | 1
Not completed — Death | 1

BASELINE CHARACTERISTICS:
Arm/Group | Experimental: Sunitinib Malate (SU011248) Treatment
Number analyzed (Participants) | 48
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 27
  >=65 years | 21
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29
  Male | 19
Region of Enrollment [Number; unit: participants]
  United States | 48

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Overall Response (OR)
Description: Objective Radiographic Response Rate. Response assessments were based on the longest diameter tumor measurements in accordance with Response Evaluation Criteria in Solid Tumors (RECIST).
Time Frame: From On Treatment to Off Study - average of 6 months
Population: All participants assessable for response
Measure: Number; unit: participants
Arm/Group | Experimental: Sunitinib Malate (SU011248) Treatment
Number analyzed (Participants) | 43
participants | 1

2. Secondary Outcome: Participants' Progression Free Survival (PFS)
Description: Time to tumor progression defined as the duration of time from start of treatment to time of progression. Response assessments were based on the longest diameter tumor measurements in accordance with Response Evaluation Criteria in Solid Tumors (RECIST).
Time Frame: From On Treatment to Off Study - average of 6 months
Population: All participants who completed the study
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Liposarcoma Cohort Only; Leiomyosarcoma Cohort Only; Malignant Fibrous Histiocytoma (MFH) Cohort Only: Experimental: Sunitinib Malate (SU011248) Treatment
Arm/Group | Liposarcoma Cohort Only | Leiomyosarcoma Cohort Only | Malignant Fibrous Histiocytoma (MFH) Cohort Only
Number analyzed (Participants) | 18 | 15 | 14
months | 3.9 [2.8 to 4.4] | 4.2 [2.0 to 8.3] | 2.5 [1.4 to 5.5]

3. Secondary Outcome: Participants' Overall Survival (OS)
Description: The median OS times (months) for liposarcoma, leiomyosarcoma and MFH.
Time Frame: From On Treatment to Off Study - average of 6 months
Population: All participants who completed the study
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Liposarcoma Cohort Only | Leiomyosarcoma Cohort Only | Malignant Fibrous Histiocytoma (MFH) Cohort Only
Number analyzed (Participants) | 18 | 15 | 14
months | 18.6 [5.2 to 27.7] | 10.1 [4.1 to 11.9] | 13.6 [3.1 to 36.5]

4. Secondary Outcome: Number of Participants With Serious Adverse Events (SAEs)
Description: Determine the number of participants who experience Serious Adverse events while on sunitinib malate study.
Time Frame: 4 years, 7 months
Population: All Participants
Measure: Number; unit: participants
Arm/Group | Experimental: Sunitinib Malate (SU011248) Treatment
Number analyzed (Participants) | 48
participants | 13

ADVERSE EVENTS:
Time Frame: 4 years, 7 months
Arm/Group | Experimental: Sunitinib Malate (SU011248) Treatment
Serious Adverse Events (participants affected / at risk) | 13/48
Other Adverse Events (participants affected / at risk) | 39/48
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Experimental: Sunitinib Malate (SU011248) Treatment (N=48)
Liver dysfunction/failure (Hepatobiliary disorders) | 1 (1)
Pain - Abdomen (General disorders) | 3 (4)
Death not associated with CTCAE term - Disease progression (General disorders) | 3 (3)
Infection with unknown ANC - Peritoneal cavity (Infections and infestations) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Cardiac general (Cardiac disorders) | 2 (2)
Hemorrhate/Bleeding (General disorders) | 2 (2)
Left ventricular systolic dysfunction (Cardiac disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Experimental: Sunitinib Malate (SU011248) Treatment (N=48)
Anorexia (Metabolism and nutrition disorders) | 10 (11)
Fatigue (General disorders) | 30 (44)
Diarrhea (Gastrointestinal disorders) | 22 (28)
Mucositis (Gastrointestinal disorders) | 18 (22)
Vomiting (Gastrointestinal disorders) | 16 (18)
Dysguesia (Gastrointestinal disorders) | 18 (24)
Dyspepsia (Gastrointestinal disorders) | 21 (22)
Thrombocytopenia (Blood and lymphatic system disorders) | 20 (27)
Neutropenia (Blood and lymphatic system disorders) | 14 (30)
Hypertension (Cardiac disorders) | 9 (9)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 7 (8)
Hemorrhage/bleeding (General disorders) | 4 (5)
Rash (Skin and subcutaneous tissue disorders) | 15 (27)

LIMITATIONS AND CAVEATS:
The trial was amended to exclude fibrosarcoma after only one patient was accrued while the other cohorts had completed 75% or more of their planned accrual. Only patients with liposarcoma, leiomyosarcoma, or MFH were enrolled after this amendment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes